CLINICAL TRIAL: NCT07360249
Title: PILOT TEST OF GLUCOSE-FRUCTOSE RATIOS ON EXOGENOUS CARBOHYDRATE OXIDATION RATES DURING EXERCISE
Brief Title: Glucose-fructose Ratio Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Professor of Nutrition and Metabolism, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11030
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Exercise Metabolism
MeSH Terms: interventions — Glucose; Fructose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One to One ratio (Experimental): Glucose and fructose ingestion in a one-to-one ratio
  Interventions: Other: Glucose and fructose (one-to-one)
- Two to one ratio (Active Comparator): Glucose and fructose ingestion in a two-to-one (1-to-0.5) ratio
  Interventions: Other: Glucose and fructose (two-to-one)

INTERVENTIONS:
Other: Glucose and fructose (one-to-one) — Glucose and fructose ingested in solution in a one-to-one ratio (135 grams per hour for 3 hours during exercise)
  Arms: One to One ratio
Other: Glucose and fructose (two-to-one) — Glucose and fructose ingested in solution in a two-to-one ratio (135 grams per hour for 3 hours during exercise)
  Arms: Two to one ratio

SUMMARY:
The aim of this pilot study is to estimate the effect size of changing the glucose-fructose ratio from 1:0.5 to 1:1 on exogenous carbohydrate oxidation rates during exercise, which can be used to power a future definitive study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above;
* Performing endurance training for at least 5 hours per week
* Capable of three hours of continuous exercise

Exclusion Criteria:

* Glucose or lipid lowering, or weight loss medication
* Diagnosis of cardiovascular disease, renal failure, liver disease or type 2 diabetes
* Contraindications to exercise
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Exogenous carbohydrate oxidation rate (g/h) | 180 minutes
  Total exogenous carbohydrate oxidation rate (g/h) over 180 minutes

SECONDARY OUTCOMES:
Peak exogenous carbohydrate oxidation rate (g/h) | 180 minutes
  Highest recorded exogenous carbohydrate oxidation rate (g/h)
Whole-body carbohydrate oxidation rate (g/h) | 180 minutes
  Total whole-body carbohydrate oxidation rate (g/h)
Endogenous carbohydrate oxidation rate (g/h) | 180 minutes
  Total endogenous carbohydrate oxidation rate (g/h)
Whole-body fat oxidation rate (g/h) | 180 minutes
  Total whole-body fat oxidation rate (g/h)
Blood lactate concentrations (mmol/L) | 180 mninutes
  Mean blood lactate concentrations over 180 minutes
Blood glucose concentrations (mmol/L) | 180 minutes
  Mean blood glucose concentrations (mmol/L) over 180 minutes
Ratings of gut comfort (arbitrary units) | 180 minutes
  Mean ratings of gut comfort (arbitrary units) over 180 minutes
Ratings of perceived exertion (arbitrary units) | 180 minutes
  Mean ratings of perceived exertion (arbitrary units) over 180 minutes

OTHER OUTCOMES:
Exogenous carbohydrate oxidation over 2 hours (g/h) | 120 minutes
  Total exogenous carbohydrate oxidation over 2 hours (g/h)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Outcome measures in anonymised format.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication in a peer-reviewed journal
Access Criteria: Via the University of Bath Research Data Repository